CLINICAL TRIAL: NCT02551822
Title: Cycling Versus Continuous Mode in Neuromodulator Programming
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: Society of Urologic Nurses and Associates (Unknown)
Responsible Party: Principal Investigator, Yuko Komesu, MD, Principal Investigator, University of New Mexico
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 12-133
Record Dates: First submitted 2015-09-09; First posted 2015-09-16 (Estimated); Results first posted 2018-04-27 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Urinary Incontinence, Urge
Keywords: Urge Urinary Incontinence, sacral neuromodulation
MeSH Terms: conditions — Urinary Incontinence, Urge

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cycling (Active Comparator): Sacral neuromodulator devices (implanted pulse generator) will be programmed to on-off cycles (on 16 seconds, off 8 seconds). This means the devices are not continuously on. Rather they are on a "cycling" program.
  Interventions: Device: sacral neuromodulator
- Continuous (Active Comparator): Sacral neuromodulator devices (implanted pulse generator) will be programmed to be on continuously. This means the devices are continuously on. They are on a "continuous" program.
  Interventions: Device: sacral neuromodulator

INTERVENTIONS:
Device: sacral neuromodulator — The Implanted Pulse Generator will be set via randomization to continuous vs cycling stimulation.
  Other Names: Interstim

SUMMARY:
The investigators objective is to compare patient outcomes as changes in validated symptom measures of overactive bladder, the Overactive Bladder Questionnaire Short Form (OABq-SF) symptom scale, between women who are set on cycling versus continuous programs for their neuromodulator. Specifically, the investigators propose to perform a randomized double blind crossover study in women who are successfully treated with neuromodulation to either continuous or cycling mode on the modulator and compare differences between groups on the validated OABq-SF symptom questionnaire. In addition, the investigators will compare differences in urinary frequency and pad counts between women randomized to cycling versus continuous stimulation as measured by a 3 day voiding diary. This investigation will provide evidence-based guidelines for neuromodulator programming.

DETAILED DESCRIPTION:
Background and Significance:

The purpose of this research proposal is to evaluate the effect of cycling versus continuous neuromodulator programming on overactive bladder syndrome. s.In 1997, the Federal Drug Administration (FDA) approved the sacral nerve stimulator as a treatment for refractory urge incontinence. Sacral Neuromodulation works via stimulation of the sacral nerve roots 2-4, (S-2, S-3 and S-4), although the exact mechanism of action is unknown. While implanted electronic stimulators have been used increasingly in the last twenty years, little investigation has documented the actual programming of the stimulator. Prospective trials examining the ideal programming parameters for a specific condition are needed to better identify optimal use of sacral nerve modulation therapy.

In brief, women with overactive bladder who are refractory to treatment are eligible for a trial placement of a neuromodulator. The modulators are placed in two stages; in stage one, a temporary lead is placed in the 3rd sacral foramen. Each neuromodulator has 4 electrodes that are placed via a single lead into the 3rd sacral foramen. The patient will generally return to clinic one week following stage 1 for a post-op evaluation. If the patient reports a 50% improvement in frequency as measured on a 3-day voiding diary, the modulator is permanently implanted. This is stage 2. After placement, the modulator is programmed in the recovery room. Patients are trialed on four set programs for their stimulator. Each program differs in electrode combination, pulse width, amplitude and rate as well as direction of current. Each of the four programs is tested with the patient to determine which is felt by the patient in the perineum and is comfortable. Finally, patients can either have their modulator set on a cycling or continuous mode. Currently, decisions regarding programming are made by whoever is assessing the patient and are not data driven.

Typically, cycling means the neuromodulator stimulation is on for 16 seconds & off for 8 seconds. Continuous means the patient receives constant stimulation. A single retrospective study described program parameters for programming of the modulator for treatment of Over Active Bladder (OAB). It described 67 patients who had good response to neuromodulation, and determined the mean pulse width was 204 microseconds, the pulse width ranged between 120-270 microseconds; the average rate was 9 with a range of 2-20 pulses/second. The majority of women were on cycling mode. Program cycling is purported to decrease the incidence of patients reporting that their modulator is no longer working and thought to extend battery life. No other study has investigated whether or not cycling of the stimulator improves patient outcomes.

Our objective is to compare patient outcomes using in validated symptom measures of OAB between women who are set on cycling versus continuous programs. Investigators propose to perform a randomized crossover study in women who are successfully treated with neuromodulation to either continuous or cycling mode and compare differences between groups on the OAB-q SF symptom questionnaire. The investigators will also compare differences in urinary frequency and pad counts between women randomized to cycling versus continuous stimulation using voiding diaries.

Specific Aims and Objectives:

Aim #1: To compare OAB improvement as measured by the Overactive Bladder Questionnaire Short Form Symptom questionnaire (OAB-q SF symptom questionnaire) between women with continuous versus cycling stimulation of their neuromodulator.

Hypothesis #1: Investigators hypothesize that women on cycling programs will report higher OAB-q SF symptom scores than women on continuous programs.

Aim #2: To compare urinary frequency as recorded on 3 day voiding diaries between women placed on continuous versus cycling stimulation of their neuromodulator.

Hypothesis #2: Investigators hypothesize that women on cycling programs report less urinary frequency as measured on 3 day voiding diaries than women on continuous programming.

Aim #3: To compare pad usage between women on cycling programs versus those on continuous programs.

Hypothesis #3: Investigators hypothesize that women on cycling programs will report less pad use than women on cycling programs.

Methods:The investigators will conduct a double-blinded crossover randomized controlled clinical trial. Up to 50 women will need to be recruited in order to randomize twenty-three women who are successful with the Stage 1 implant of their neuromodulator. After written consent, clinical data will be collected and questionnaires administered. After successful Stage 1 placement women will complete a 3-day voiding diary. The recording of symptoms and completion of a voiding diary are standard of care for women undergoing neuromodulation treatment. These data will be collected and recorded.

Randomization will occur after successful Stage 2 implantation. Study personnel not otherwise involved in patient care will assign it. Randomization assignment will be by random number table in permutated blocks of four, to ensure that equal numbers of women will be assigned to each group. Assignments will be kept in sealed opaque envelopes and will be opened in sequential order once women have undergone successful Stage 2 implantation. Study personnel programming the modulator after implantation will either program the modulator to continuous or cycling programs. Patients will be blinded to randomization assignment.

Prior to their 3 month visit, study subjects will complete another voiding diary. At the visit, women will complete the OAB-q SF symptom questionnaire as well as the Patient Global Impression of Improvement (PGI-I). At this visit, women who were assigned to continuous stimulation will be switched to cycling stimulation and women who were assigned to cycling stimulation will be switched to continuous stimulation. Women again will report for clinical follow-up at six months. Women will be asked to complete their voiding diary. At this clinic visit women will once again complete the OAB-q SF symptoms questionnaire and PGI-I

Investigators obtain a written consent from qualifying patient. Patients will then be randomized to Cycling or Continuous mode at Stage II implantation.

Statistics:

Analysis: Descriptive statistics will be used to describe patient characteristics. The analysis of the change in OAB-q SF scores in this 2 group, 2 period (2x2) crossover design will be a repeated measures (RM) Analyses of Variance (ANOVA) with both the treatment group (cycling versus continuous) and period (first treatment versus second treatment) as repeated factors. The possibility of a cross over effect will be accounted for in the analysis by an order effect covariate (equal to 1 if cycling is first and 0 if not.) Analysis of urinary incontinence episodes and pad counts as recorded on 3 day voiding diaries will be analyzed by repeated measures Poisson regression. (Using SAS's PROC GEN MOD with a Poisson distribution) Significance is set at p = 0.05.

Power analysis: In our cross over randomized controlled trial the investigators assume that a clinically important difference between changes in OAB-q SF scores between women on continuous versus cycling stimulation, with a standard deviation of the paired differences of 15 points between groups with an alpha error of 0.05 and power of 80%, 20 women are needed to be randomized into equal groups.

(Hintze, J (2011) PASS11. NCSS, LLC< Kaysville Utah, US. www.ncss.com)(9), Assuming that 15% of women will be lost to follow-up the investigators will need to randomize 23 women to the study.

2. Expected outcome: This randomized control trial will demonstrate that women on the cycling program mode will report higher OAB-q SF Symptom scores, and will report less urinary frequency and less pad usage as measured on 3-day voiding diaries.

ELIGIBILITY:
Inclusion Criteria:

* Women at least 21 years old or older eligible for implantation of a neuromodulator
* Women with successful Stage #1 implantation for treatment of refractory OAB
* Subjects may be enrolled in other studies as long as there are no changes to the neuromodulation device. Women may continue other OAB therapies that they are on, but as asked to not start new therapies.
* Not currently pregnant and with no plans to become pregnant during the course of the trial.
* Willing as well as mentally and physically capable of completing all study related procedures and materials

Exclusion Criteria:

* Males (we do not care for males in our urogynecology clinic)
* Incarcerated women
* Non-English speakers
* Pregnant women
* Scheduled or planned MRIs or diathermy

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuko M Komesu, MD, Principal Investigator — University of New Mexico Health Sciences Center; Gwendolyn Beer, RN, Study Chair — University of New Mexico Health Sciences Center; Rebecca G Rogers, MD, Study Director — University of New Mexico Health Sciences Center
Locations (2):
- United States (2):
  - University of New Mexico Hospital, Albuquerque, New Mexico
  - University of New Mexico Health Science Center, Albuquerque, New Mexico

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 9 participants were withdrawn or lost to follow-up prior to randomization. 32 participants enrolled and 23 were randomized.
Groups:
- Cycling, Then Continuous; Continuous, Then Cycling: Women will be randomized to the continuing or cycling arm at 0 months. At 3 months, women will report for their second postoperative visit. Prior to this visit, study subjects will complete the third 3-day voiding diary and record pad usage. At the visit, women will complete the OAB-q SF as well as the PGI-I, and will be queried regarding any complications since the start of the use of their modulator. At the 3 month visit, women who were assigned to continuous stimulation will be switched to cycling stimulation and women who were assigned to cycling stimulation will be switched to continuous stimulation. Women again will report for clinical follow-up at six months. Women will be asked to complete a fourth 3 day voiding diary. In addition, women will be asked to record any complications that they have had in the preceding 3 months. At this clinic visit women will once again complete the OAB-q SF and PGI-I.
Period: Overall Study
Arm/Group | Cycling, Then Continuous | Continuous, Then Cycling
Started | 11 | 12
Completed | 9 | 10
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Group A (Cycling, Then Continuous): Sacral neuromodulator devices (implanted pulse generator) will be programmed to on-off cycles (on 16 seconds, off 8 seconds). This means the devices are not continuously on. Rather they are on a "cycling" program.
  sacral neuromodulator: The Implanted Pulse Generator will be set via randomization to continuous vs cycling stimulation.
  The first intervention (cycling) occurred at baseline, and the second intervention occurred at 3 months (continuous).
- Group B (Continuous, Then Cycling): Sacral neuromodulator devices (implanted pulse generator) will be programmed to be on continuously. This means the devices are continuously on. They are on a "continuous" program.
  sacral neuromodulator: The Implanted Pulse Generator will be set via randomization to continuous vs cycling stimulation.
  The first intervention (continuous) occurred at baseline, and the second intervention occurred at 3 months (cycling).
- Total: Total of all reporting groups
Arm/Group | Group A (Cycling, Then Continuous) | Group B (Continuous, Then Cycling) | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.8 (10.4) | 63.4 (13.1) | 66.5 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic Latina | 5 | 5 | 10
  White | 6 | 2 | 8
  Black | 0 | 3 | 3
  American Indian | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Overactive Bladder Questionnaire-Short Form (OABq) Short Form Symptom Bother Scale Result
Description: The Overactive Bladder Questionnaire (OAB-q) assesses symptom bother & health-related quality of life (HRQL) for overactive bladder. The short form OAB-q SF, provides a quick assessment of symptom bother, consisting of a 6-item symptom bother scale. The questionnaire is on a 6 point scale, 1 indicates symptom is not bothersome (best outcome), 6 indicates symptom bothers the participant "a very great deal" (worst possible outcome). The majority of the participants were missing the HRQL portion of the questionnaire, so this portion of the questionnaire was not included in the analysis. These are the raw scores ranges for each question prior to being transformed. The possible scores for complete surveys range from 13 (if the participant marked "not bothersome" for all 6) to 78 (if the participant marked "a very great deal" for all 6 questions) once transformed. The reported numbers are the transformed scores [(actual raw score-lowest possible score)/possible raw score range] X 100.
Time Frame: Three months after change in program from cycling to continuous or vice versa.
Population: Two participants in group A and two participants in group B withdrew from the study prior to completion.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Cycling, Then Continuous: Sacral neuromodulator devices (implanted pulse generator) will be programmed to on-off cycles (on 16 seconds, off 8 seconds). This means the devices are not continuously on. Rather they are on a "cycling" program.
  sacral neuromodulator: The Implanted Pulse Generator will be set via randomization to continuous vs cycling stimulation.
- Continuous, Then Cycling: Sacral neuromodulator devices (implanted pulse generator) will be programmed to be on continuously. This means the devices are continuously on. They are on a "continuous" program.
  sacral neuromodulator: The Implanted Pulse Generator will be set via randomization to continuous vs cycling stimulation.
Arm/Group | Cycling, Then Continuous | Continuous, Then Cycling
Number analyzed (Participants) | 11 | 12
units on a scale
  Baseline | 68.3 (22.3) | 66.3 (27.0)
  3 Months: number analyzed (Participants) | 10 | 12
  3 Months | 30.3 (20.7) | 38.0 (22.0)
  6 Months: number analyzed (Participants) | 09 | 10
  6 Months | 24.7 (20.7) | 53.3 (27.0)

2. Secondary Outcome: Voiding Diary: Urge Incontinence Episodes
Description: Bladder Diaries (BD) are a useful clinical tool and one of the most common outcome measure used in studies of urinary incontinence and other forms of lower urinary tract dysfunction. The patient is asked to prospectively record the frequency, number and volume of voids and incontinence episodes. The National Institutes of Health (NIH) recommends diary duration of at least three days for research studies.
Time Frame: Three months after change in program from cycling to continuous or vice versa.
Population: 2 Participants from group A and two participants from group B withdrew from the study prior to completion.
Measure: Mean (Standard Deviation); unit: Number of leaks per day on 3 day diary
Arm/Group | Cycling, Then Continuous | Continuous, Then Cycling
Number analyzed (Participants) | 11 | 12
Number of leaks per day on 3 day diary
  Baseline | 6.9 (3.4) | 8.1 (6.5)
  Change to 3 Months: number analyzed (Participants) | 10 | 12
  Change to 3 Months | -1.3 (4.5) | -2.9 (7.4)
  Change to 6 Months: number analyzed (Participants) | 09 | 10
  Change to 6 Months | -.35 (5.7) | -2.5 (6.3)

3. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) Questionnaire Scale Results
Description: The Patient Global Impression of Improvement (PGI-I) scale is a global index that may be used to rate the response of a condition to a therapy. It is a transition scale that is a single question asking the patient to rate their urinary tract condition now, as compared with how it was prior to before beginning treatment on a 7 point scale, 1 indicating the participant's condition is "Very much better" (best possible outcome), and 7 being "Very much worse" (worst possible outcome). The answers to the 7 questions were then averaged to a score.
Time Frame: Three months after change in program from cycling to continuous or vice versa.
Population: 2 Participants in group A and 2 participants in group B withdrew from the study prior to completion.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cycling, Then Continuous | Continuous, Then Cycling
Number analyzed (Participants) | 11 | 12
units on a scale
  3 Months: number analyzed (Participants) | 10 | 12
  3 Months | 2.6 (1.3) | 2.6 (.79)
  6 Months: number analyzed (Participants) | 09 | 10
  6 Months | 2.5 (1.5) | 2.7 (1.7)

ADVERSE EVENTS:
Groups:
- Arm 1: Cycling: Sacral neuromodulator devices (implanted pulse generator) will be programmed to on-off cycles (on 16 seconds, off 8 seconds). This means the devices are not continuously on. Rather they are on a "cycling" program.
  sacral neuromodulator: The Implanted Pulse Generator will be set via randomization to continuous vs cycling stimulation.
- Arm 2: Continuous: Sacral neuromodulator devices (implanted pulse generator) will be programmed to be on continuously. This means the devices are continuously on. They are on a "continuous" program.
  sacral neuromodulator: The Implanted Pulse Generator will be set via randomization to continuous vs cycling stimulation.
Arm/Group | Arm 1: Cycling | Arm 2: Continuous
All-Cause Mortality (participants affected / at risk) | 1/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 1/23
Other Adverse Events (participants affected / at risk) | 8/23 | 9/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Cycling (N=23) | Arm 2: Continuous (N=23)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) — The Participant had a history of seizures, and one occurred during study participation. The participant did not go to the hospital.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Cycling (N=23) | Arm 2: Continuous (N=23)
Falls (Injury, poisoning and procedural complications) | 5 | 4
Current Urinary Tract Infection (Infections and infestations) | 1 | 2 — The participant in group A received antibiotics. One out of the two participants in group B received antibiotics. All instances of UTIs occurred at 6 months post implant.
Changes in bowel movements (Gastrointestinal disorders) | 2 | 4 — Symptoms include constipation, diarrhea, both, or other.
New Treatments for OAB (Renal and urinary disorders) | 2 | 1
Stopped medications for OAB (Renal and urinary disorders) | 0 | 2
Outpatient Surgery (Surgical and medical procedures) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No